CLINICAL TRIAL: NCT03363659
Title: A Phase II, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Disulfiram and Copper Gluconate When Added to Standard Temozolomide Treatment in Patients With Newly Diagnosed Resected Unmethylated Glioblastoma Multiforme
Brief Title: Disulfiram and Copper Gluconate With Temozolomide in Unmethylated Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17.56
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
Keywords: Glioblastoma; Glioblastoma Multiforme; Anaplastic Glioma; Unmethylated
MeSH Terms: conditions — Glioblastoma | interventions — Disulfiram; Gluconates; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DSF-Cu with temozolomide and radiation (Experimental): Disulfiram (DSF; oral) / copper gluconate (Cu; oral) dosed at 125 mg / 2 mg, twice daily. Temozolomide will be administered following the standard Stupp protocol at a dose of 75 mg/m2 for 42 days with concurrent radiation therapy. Temozolomide maintenance dose will be 150 mg/m2 once daily on Days 1-5 of every 28-day cycle while DSF-Cu is continued twice daily, as tolerated, for the duration of the Temozolomide adjuvant treatment. Patients demonstrating continued benefit from the adjuvant temozolomide after 6 cycles can continue treatment to a maximum of 12 cycles
  Interventions: Drug: Disulfiram; Dietary Supplement: Copper gluconate; Drug: Temozolomide

INTERVENTIONS:
Drug: Disulfiram — Disulfiram is taken orally, twice daily.
  Other Names: Antabuse
Dietary Supplement: Copper gluconate — Copper gluconate is taken orally, twice daily
Drug: Temozolomide — Temozolomide is taken once daily
  Other Names: Temodar, Temodal, Temcad

SUMMARY:
One of Disulfiram antitumor effects suggested in preclinical studies is MGMT (methyl-guanine-methyl-transferase) inhibition. Disulfiram MGMT inhibitory effect is enhanced by addition of Copper. This study evaluates the impact of Disulfiram (DSF) + Copper (Cu) combination when added to standard Temozolomide in the treatment of unmethylated Glioblastoma Multiforme (GBM) patients.

DETAILED DESCRIPTION:
Glioblastoma is the most common malignant primary brain tumor and one of the most devastating cancers. The current standard of care for glioblastoma includes maximal safe resection followed by radiotherapy and temozolomide, which results in a median progression-free survival of less than 7 months, and median overall survival (OS) of less than 15 months. Moreover, patients with unmethylated glioblastoma respond poorly to this current standard treatment. This clinical trial evaluates the potential role of continuous, upfront use of Disulfiram in combination with Copper gluconate in enhancing temozolomide effect in the treatment of unmethylated Glioblastoma multiforme (GBM) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of histologically confirmed glioblastoma (WHO grade IV). Subjects with an original histologic diagnosis of low grade glioma or anaplastic glioma (WHO grade II or III) are eligible if a subsequent histological diagnosis of glioblastoma is made
* Patients whose tumor is determined to be unmethylated
* Patients with incomplete resection as determined by residual, measurable gadolinium or contrast-enhancing lesion or lesions
* Recent resection of glioblastoma within 4 weeks of study entry. Patients who have only had a tumor biopsy and who are considered unresectable are eligible (but based on the study accrual this subset of patients with unresectable tumor may be considered for separate analysis)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of ≤ 2 (see appendix A)
* Willing to remain abstinent from consuming alcohol while on DSF
* No prior radiation or chemotherapy
* Meets the following laboratory criteria:

  * Absolute neutrophil count ≥ 1,500/mcL (microliter)
  * Platelets ≥ 100,000/mcL
  * Hemoglobin > 10.0 g/dL (grams/deciliter) (transfusion and/or ESA (erythropoiesis-stimulating agent) allowed)
  * Total bilirubin and alkaline phosphatase ≤ 2x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
  * Blood urea nitrogen (BUN) and creatinine < 1.5 x ULN
* Able to take oral medication
* Able to understand and willing to sign an institutional review board (IRB)-approved written informed consent document (legally authorized representative permitted)

Exclusion Criteria:

* Radiographic evidence of leptomeningeal dissemination, extensive intraparenchymal dissemination, infratentorial tumor, or metastatic disease to sites remote from the supratentorial brain
* Enrolled in another clinical trial testing a novel therapy or drug
* Received prior radiation therapy or chemotherapy for glioblastoma
* History of allergic reaction/hypersensitivity to DSF (without alcohol) or copper.
* Treatment with the following medications that may interfere with metabolism of DSF: warfarin (unless otherwise chosen by the study PI who will actively adjust Coumadin dose to consistently maintain a safe, therapeutic international normalized ratio (INR) < 3, theophylline, amitriptyline, isoniazid, metronidazole, phenytoin, phenobarbital, chlorzoxazone, halothane, imipramine, chlordiazepoxide, diazepam. (Note: lorazepam and oxazepam are not affected by the P450 system and are not contraindicated with DSF).
* Active severe hepatic or renal disease
* Grade 2 or higher peripheral neuropathy or ataxia per NCI CTCAE version 4.0 (2009)
* History of idiopathic seizure disorder schizophrenia, or psychosis unrelated to glioblastoma, corticosteroid, or anti-epileptic medications
* History of Wilson's or Gilbert's disease
* Current excessive use of alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asadullah Khan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrollment 28th March 2018. Subjects screened at neuro-oncology MDCC (Multi-disciplinary cancer clinic) and enrolled at neuro-oncology clinic.
  Study closed 13th January 2022.
Groups:
- Open Label: Open-Label, Single Arm Study to Evaluate the Safety, Tolerability, and Efficacy of Disulfiram and Copper Gluconate When Added to Standard Temozolomide Treatment in Patients with Newly Diagnosed Resected Unmethylated Glioblastoma Multiforme
Period: Overall Study
Arm/Group | Open Label
Started | 15 (Of 15 subjects consented, 1 subject was a screen fail and 1 subject withdrew before any planned intervention.)
Completed | 12
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Screen fail | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 15 subjects consented, 1 subject was a screen fail and 1 subject withdrew before any planned intervention.
Groups:
- Open Label: Open-Label, Single Arm Study to Evaluate the Safety, Tolerability, and Efficacy of Disulfiram and Copper Gluconate When Added to Standard Temozolomide Treatment in Patients with Newly Diagnosed Resected Unmethylated Glioblastoma Multiforme.
  DSF will be given at 125 mg (half of a 250 mg capsule) two times daily with meals. Cu gluconate will be taken with each dose of DSF at a dose of 2 mg (one capsule/tablet). The DSF total daily dose will be 250 mg per day, as lower dose may be associated with a higher MGMT inhibitory effect.
Arm/Group | Open Label
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: 15 subjects consented, Age data was not collected for 2 participants - 1 subject was a screen fail and 1 subject withdrew before any planned intervention.
  Participants
    number analyzed (Participants) | 13
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Both men and women and members of all races and ethnic groups are eligible for this trial
  Participants
    Female | 3
    Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: 6 Months Progression Free Survival (PFS)
Description: To determine 6 month PFS of patients with unmethylated glioblastoma treated with DSF-Cu in combination with concurrent radiation and temozolomide. This was assessed by the number of participants who did not have disease progression and were alive at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 12
Participants | 1

2. Primary Outcome: Overall Survival
Description: Overall Survival will be assessed as a number of participants alive at 1 and 2 years.
Time Frame: 1 and 2 years
Population: 2 participants are not included here because 1 was a screen fail and 1 withdrew before starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 13
Participants
  1 Year | 9
  2 Years | 2

3. Secondary Outcome: Quality of Life (QOL)
Description: Edmonton Symptom Assessment System - Revised (ESAS-r) questionnaire
Time Frame: 1 year
Population: Disease progression or required dose modification from all participants took them all off the study. No data was collected.
Arm/Group | Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Reportable adverse events will be tracked for 30 days after the last dose of DSF-Cu. Survival for participants was followed for up to 2 years.
Description: 13 participants started the treatment and the only ones assessed for adverse events. All participants were included in all cause mortality.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 11/15
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=13)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) — 60 year old female with a history of Glioblastoma multiforme, presented with increased fatigue and new onset jaundice. Liver biopsy, which favored drug-induced liver injury likely due to chemotherapy agents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT03363659/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03363659/ICF_001.pdf